CLINICAL TRIAL: NCT00101335
Title: A Phase IIb Cancer Prevention Trial of Celecoxib, a Selective COX-2 Inhibitor, in Oral Leukoplakia
Brief Title: Celecoxib in Preventing Head and Neck Cancer in Patients With Oral Leukoplakia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Fox Chase Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Masking: Double | Purpose: Prevention
Other Study IDs: FCCC-02028; CDR0000393574 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2005-01-07; First posted 2005-01-10 (Estimated); Last update posted 2013-07-11 (Estimated); Status verified 2013-07

CONDITIONS: Head and Neck Cancer; Precancerous Condition
Keywords: hypopharyngeal cancer; lip and oral cavity cancer; nasopharyngeal cancer; oropharyngeal cancer; tongue cancer; oral leukoplakia
MeSH Terms: conditions — Head and Neck Neoplasms; Precancerous Conditions; Hypopharyngeal Neoplasms; Mouth Neoplasms; Nasopharyngeal Neoplasms; Oropharyngeal Neoplasms; Tongue Neoplasms; Leukoplakia, Oral | interventions — Celecoxib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: celecoxib

SUMMARY:
RATIONALE: Chemoprevention is the use of certain drugs to keep cancer from forming, growing, or coming back. The use of celecoxib may prevent or treat head and neck cancer.

PURPOSE: This randomized phase II trial is studying celecoxib to see how well it works compared to placebo in preventing head and neck cancer in patients with oral leukoplakia.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Compare the clinical efficacy of celecoxib vs placebo, in terms of inducing regression of oral leukoplakia lesions, in patients with hyperplastic or dysplastic oral leukoplakia.

Secondary

* Determine the effect of this drug in modulating multiple intermediate biomarkers (e.g., COX-2, PPARγ, or PPARδ) in normal and hyperplastic or dysplastic oral epithelia of these patients.
* Determine the safety of this drug in these patients.
* Determine the cost-effectiveness of this drug as a chemopreventative agent in these patients.

OUTLINE: This is a randomized, double-blind, placebo-controlled, cross-over study. Patients are stratified according to the pathology of the leukoplakia lesion (dysplasia vs hyperplasia). Patients are randomized to 1 of 2 arms.

* Arm I: Patients receive oral celecoxib twice daily for 3 months.
* Arm II: Patients receive oral placebo twice daily for 3 months. All patients undergo biopsy. Patients then cross-over to the opposite treatment arm for 3 months.

In both arms, treatment continues in the absence of unacceptable toxicity or disease progression.

Patients are followed at 1 month.

PROJECTED ACCRUAL: A total of 27-60 patients (18-40 for study drug, 9-20 for placebo before cross-over) will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of oral leukoplakia with hyperplasia or dysplasia

  * Documented by baseline biopsy of oral lesions suspicious for leukoplakia
  * For patients using dentures over the past 6 months, only lesions located on the ventral-lateral tongue or floor of the mouth are allowed
  * No leukoplakia/hyperplasia secondary to mechanical irritation
* No carcinoma in situ of the oral cavity

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* Not specified

Life expectancy

* At least 1 year

Hematopoietic

* Hemoglobin ≥ 10 g/dL (women) OR ≥ 11 g/dL (men)

Hepatic

* AST or ALT normal
* Bilirubin normal

Renal

* Creatinine normal OR
* Creatinine clearance ≥ 60 mL/min

Cardiovascular

* No myocardial infarction within the past 12 months
* No known active ischemic cardiac disease by stress test or echocardiogram

Gastrointestinal

* No history of gastrointestinal hemorrhage
* No known gastrointestinal ulcers within the past 2 years unless there is documentation of healed lesions by upper endoscopy
* No active or suspected peptic ulcer disease
* Negative stool guaiac test

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 2 months after study treatment
* No use of snuff or chewing tobacco within the past 2 months
* No active invasive malignancy within the past 3 years except nonmelanoma skin cancer or in situ carcinomas
* No clinical evidence of chronic infectious disease
* No clinical evidence of connective tissue disease
* No known hypersensitivity (asthma, urticaria, or acute rhinitis induced by NSAIDs) to aspirin or other NSAIDs
* No known hypersensitivity to sulfonamides

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* Not specified

Endocrine therapy

* At least 6 months since prior chronic or frequent use of systemic glucocorticoids
* No concurrent chronic or frequent use of systemic glucocorticoids

Radiotherapy

* Not specified

Surgery

* Not specified

Other

* No prior chronic or frequent (> 100 mg per day aspirin equivalent) use of nonsteroidal anti-inflammatory drugs (NSAIDs) for 7 of the past 14 days
* At least 3 months since prior experimental therapy
* No concurrent chronic or frequent use of NSAIDs

  * Cardioprotective doses of aspirin ≤ 100 mg daily are allowed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2003-11; Primary Completion 2005-01 (Actual); Study Completion 2005-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul F. Engstrom, MD, Principal Investigator — Fox Chase Cancer Center
Locations (1):
- Fox Chase Cancer Center, Philadelphia, Pennsylvania, United States